CLINICAL TRIAL: NCT00014378
Title: A Phase I Study Of The Chinese Herb Huanglian (Coptis Chinesis) In Patients With Advanced Solid Tumors
Brief Title: Huang Lian (Chinese Herb) in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-061; MSKCC-00061; NCI-H01-0069
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Coptidis rhizoma extract

ARMS (1):
- Chinese Herb Huanglian (Coptis chinesis) (Experimental)
  Interventions: Drug: Chinese Herb Huanglian (Coptis chinesis)

INTERVENTIONS:
Drug: Chinese Herb Huanglian (Coptis chinesis) — Patients will receive capsules of the powdered extract of the huanglian root, which will take by mouth 4 times a day (qid).

SUMMARY:
RATIONALE: The Chinese herb Huang Lian contains ingredients that may slow the growth of cancer cells and may be an effective treatment for solid tumors.

PURPOSE: Phase I trial to study the effectiveness of Huang Lian in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of Huang Lian (Chinese herb) in patients with advanced solid tumors.
* Determine the optimal pharmacologic, molecular, and biologic parameters of this treatment regimen in these patients.
* Assess the preliminary therapeutic activity of this treatment regimen in this patient population.

OUTLINE: This is a dose-escalation study.

Patients receive oral Huang Lian (Chinese herb) 4 times daily. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of Huang Lian until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-liming toxicity.

PROJECTED ACCRUAL: Approximately 20-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor refractory to standard therapy or for which no standard therapy exists
* Measurable or evaluable disease
* No CNS primary tumor or metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,500/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No history of cardiac arrhythmias (including atrial fibrillation)
* No congestive heart failure
* No angina or myocardial infarction within the past 6 months
* QTc interval no greater than 0.48 sec

Other:

* Potassium at least 3.5 mEq/L
* Magnesium at least 1.4 mEq/L
* No mental incapacity that would preclude informed consent
* No serious or uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* At least 2 weeks since prior herbal therapy for cancer and recovered
* No concurrent class IA or III antiarrhythmic agents (e.g., quinidine, procainamide, disopyramide, sotalol, amiodarone, ibutilide, almokalant, or dofetilide)
* No concurrent tricyclic antidepressants (e.g., amitriptyline, doxepin, desipramine, imipramine, or clomipramine)
* No concurrent antiseizure medication (including dilantin and phenobarbital) for any underlying seizure disorder

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2000-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States